CLINICAL TRIAL: NCT01493622
Title: A Double-Blind,Randomized Study of Minocycline for the Treatment of Negative and Cognitive Symptoms in Schizophrenia
Brief Title: The Study of Minocycline for Negative and Cognitive Symptoms in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Fang Liu, Mental Health Institute of the Second Xiangya Hospital, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSU-2010-PSY; 2010LL02 (Other: The First Affiliated Hospital of Kunming Medical College)
Record Dates: First submitted 2010-12-20; First posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia minocycline cognition
MeSH Terms: conditions — Schizophrenia | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Subjects will be given with 200mg/day placebo(100mg,bid) and variable dose SGA. All drugs will be administered orally.
  Interventions: Drug: placebo
- minocycline (Active Comparator): Subjects will be given with 200mg/day minocycline (100mg,bid)and variable dose SGA.All drugs will be administered orally.
  Interventions: Drug: minocycline

INTERVENTIONS:
Drug: minocycline — variable dose SGA and minocycline,100mg per capsule po（take orally） bid，16 weeks；
  Other Names: Minocycline Hydrochloride Capsules
  Arms: minocycline
Drug: placebo — variable dose SGA and 100mg per capsule po（take orally） bid，16 weeks；
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether minocycline are effective in the treatment of negative and cognitive symptoms in schizophrenia.

DETAILED DESCRIPTION:
Immune-related disorders have been hypothesized as etiological factors in schizophrenia.Minocycline is a second-generation tetracycline that exerts anti-inflammatory and antimicrobial effects while having a distinct neuroprotective profile.This study was performed as a double-blind, placebocontrolled,randomized evaluation of Second generation antipsychotics(SGA) and minocycline versus SGA and placebo.

ELIGIBILITY:
Inclusion Criteria:

* male and female,were aged 18-40 years
* were currently diagnosed with DSM-IV schizophrenia
* were able to comprehend the cognition test
* patients or guardian signed informed consent,were able to comprehend the procedure and aims of the study,agreed to join the study
* patient's current antipsychotic medication regimen must be stable
* must be in a stable living arrangement

Exclusion Criteria:

* had ever been hypersensitivity to minocycline or tetracycline;
* had acute,unstable,significant,or untreated medical illness besides schizophrenia
* were pregnant or breast-feeding;
* had a DSM-IV diagnosis of substance abuse or dependency;
* had a tendency to suicide or Violence,self-harm;
* had taken immunosuppressive agents in the preceding 3 months before study entry;
* had influenza or fever in the preceding 2 weeks before study entry;
* had a DSM-IV diagnosis of emotional psychosis,Mental retardation,etc.
* has suicidal attempts or ideation or violent behavior within the last 12 months
* patient has mental retardation or severe organic brain syndromes
* treatment with Electroconvulsive Therapy (ECT) within 6 months prior to screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in the Composite Score From the Cognition Assessment Battery and SANS Total Scores After 16 Weeks of Treatment | 16 weeks
  The Cognitive Assessment Battery included Making Test (TMT) ,Symbol Coding,Hopkins Verbal Learning Test-Revised ,Mazes,Brief Visuospatial Memory Test-Revised ,Continuous Performance Test-Identical Pairs,Grooved Pegboard Test,Color Trail Test,Stroop Task,Verbal Fluency,Paced Auditory Serial Addition Test and Wisconsin Card Sorting Test SANS=Scale for the Assessment of Negative Symptoms

SECONDARY OUTCOMES:
Mean Change from Baseline in the PANSS and PSP Total Scores after 16 weeks Treatment | 16 weeks
Cytokine Measure | 16 weeks
  Cytokine Measure:IL-1β,IL-6,TNF-α,Nitric Oxide (NO)、S100B
metabolic index | 16 weeks
  weight,height,insulin and waist circumference,

CONTACTS AND LOCATIONS:
Overall Officials: Zhao J Ping, Principal Investigator — The Second Xiangya Hospital, Central South University,China
Locations (1):
- Department of Psychiatry, The First Affiliated Hospital of Kunming Medical College, Kunming, Yunnan, China

REFERENCES:
- [Result] Levkovitz Y, Mendlovich S, Riwkes S, Braw Y, Levkovitch-Verbin H, Gal G, Fennig S, Treves I, Kron S. A double-blind, randomized study of minocycline for the treatment of negative and cognitive symptoms in early-phase schizophrenia. J Clin Psychiatry. 2010 Feb;71(2):138-49. doi: 10.4088/JCP.08m04666yel. Epub 2009 Nov 3. PMID 19895780
- [Derived] Liu F, Zhang B, Xie L, Ruan Y, Xu X, Zeng Y, Messina L, Zhao J, Fan X. Changes in plasma levels of nitric oxide metabolites and negative symptoms after 16-week minocycline treatment in patients with schizophrenia. Schizophr Res. 2018 Sep;199:390-394. doi: 10.1016/j.schres.2018.03.003. Epub 2018 Mar 9. PMID 29526457
- [Derived] Liu F, Guo X, Wu R, Ou J, Zheng Y, Zhang B, Xie L, Zhang L, Yang L, Yang S, Yang J, Ruan Y, Zeng Y, Xu X, Zhao J. Minocycline supplementation for treatment of negative symptoms in early-phase schizophrenia: a double blind, randomized, controlled trial. Schizophr Res. 2014 Mar;153(1-3):169-76. doi: 10.1016/j.schres.2014.01.011. Epub 2014 Feb 3. PMID 24503176